CLINICAL TRIAL: NCT01653678
Title: Effect of Vitamin D and Omega-3 Fatty Acids on Blood Pressure and Hypertension
Brief Title: Vitamin D and Omega-3 Hypertension Trial (VITAL Hypertension)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Howard D. Sesso, ScD, MPH, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2010-P-002880; 1R01HL102122 (NIH)
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hypertension
Keywords: vitamin D-3; omega-3 fatty acids; fish oil; hypertension; blood pressure
MeSH Terms: conditions — Hypertension | interventions — Cholecalciferol; Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin D + fish oil (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D-3 (cholecalciferol), 2000 IU; Drug: Omega-3 fatty acids (fish oil)
- Vitamin D + fish oil placebo (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D-3 (cholecalciferol), 2000 IU; Drug: Fish oil placebo
- Vitamin D placebo + fish oil (Active Comparator)
  Interventions: Drug: Omega-3 fatty acids (fish oil); Dietary Supplement: Vitamin D placebo
- Vitamin D placebo + fish oil placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Vitamin D placebo; Drug: Fish oil placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D-3 (cholecalciferol), 2000 IU
  Other Names: cholecalciferol
  Arms: Vitamin D + fish oil; Vitamin D + fish oil placebo
Drug: Omega-3 fatty acids (fish oil) — Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Arms: Vitamin D + fish oil; Vitamin D placebo + fish oil
Dietary Supplement: Vitamin D placebo
  Arms: Vitamin D placebo + fish oil; Vitamin D placebo + fish oil placebo
Drug: Fish oil placebo
  Arms: Vitamin D + fish oil placebo; Vitamin D placebo + fish oil placebo

SUMMARY:
The VITamin D and OmegA-3 TriaL (VITAL; NCT 01169259) is an ongoing randomized clinical trial in 25,875 U.S. men and women investigating whether taking daily dietary supplements of vitamin D3 (2000 IU) or omega-3 fatty acids (Omacor® fish oil, 1 gram) reduces the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses. The VITAL Hypertension ancillary study is being conducted among participants in VITAL and will examine whether vitamin D or omega-3 fatty acids are related to changes in blood pressure and hypertension.

DETAILED DESCRIPTION:
The human toll of hypertension is staggering, and effective preventive measures are needed. Studies suggest that inadequate vitamin D and omega-3 fatty acid levels may be involved in the development of hypertension through multiple pathways. Results from several small clinical trials suggest that these agents may have blood pressure lowering effects, however, larger trials using higher doses of both vitamin D and omega-3 fatty acids for the prevention of hypertension among people with normal blood pressure levels are lacking. The VITamin D and OmegA-3 TriaL (VITAL) provides a cost-effective setting to examine the effects of both study agents on changes in blood pressure and new diagnoses of hypertension.

VITAL Hypertension will test the following hypotheses: (1) whether vitamin D and fish oil supplementation lowers 24-hour blood ambulatory blood pressure (ABP) compared to placebo in a subcohort of 1,000 participants; (2) whether vitamin D and fish oil supplementation reduces the risk of incident hypertension compared to placebo among all randomized VITAL participants without baseline hypertension; and (3) whether vitamin D and fish oil supplementation favorably change hypertension-related biomarkers that are potential mechanisms linking vitamin D and omega-3 fatty acids with hypertension compared to placebo.

A representative subcohort of 1,000 VITAL participants without hypertension from selected major metropolitan areas throughout the US will be invited to participate in home-based study visits at baseline and 2 years follow-up. During these visits, participants will be asked to wear monitors to record 24-hour ABP measurements, provide fasting bloods, spot urine samples, and other clinical measurements. The visits will be conducted by Examination Management Services, Inc. (EMSI), a nationally based, clinical services provider. We will compare 2-year changes in ABP among those randomized to vitamin D and omega-3 fatty acid supplements versus those randomized to placebo. In addition, we will assess the 2-year changes in levels of clinically and mechanistically relevant biomarkers of hypertension compared the 2 treatment groups.

New diagnoses of hypertension among all VITAL participants will be ascertained on annual follow-up questionnaires. To strengthen our classification of hypertension status, we will supplement our questionnaire data with annual updates of hypertension information based upon outpatient diagnostic codes and medication prescription usage from the Centers for Medicare & Medicaid Services (CMS) database. Incidence of hypertension among those assigned to each active agent versus placebo will be compared.

In addition, baseline blood samples from 1,000 participants with new diagnoses of hypertension will be compared with those from 2,000 participants without hypertension to determine whether the effect of vitamin D and/or omega-3 fatty acid supplements on the incidence of hypertension is modified by baseline plasma levels of vitamin D or omega-3 fatty acids.

Results from VITAL Hypertension will provide important evidence to support or refute the potential preventive roles of vitamin D and omega-3 fatty acids on blood pressure and the development of hypertension.

ELIGIBILITY:
Participants eligible and willing to participate in the main VITAL trial (NCT 01169259) who meet the following criteria are eligible to participate in the VITAL Hypertension ancillary study: all participants with no baseline history of hypertension and, for home visits in the subcohort of 1,000 participants, those living in selected cities throughout the U.S..

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25875 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2025-11 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure | Two years
  Change in 24-hour ambulatory blood pressure measurements among a subcohort of approximately 1,000 participants.
Incident hypertension | 5 years
  Incidence of hypertension in the overall VITAL trial cohort.
Changes in 25-hydroxy-vitamin D levels | 2 years
  Changes in a subcohort of approximately 1,000 participants.
Changes in fatty acid levels | 2 years
  Changes in a subcohort of approximately 1,000 participants
Changes in biomarkers related to blood pressure | 2 years
  Changes in a subcohort of approximately 1,000 participants

CONTACTS AND LOCATIONS:
Overall Officials: Howard D. Sesso, ScD, MPH, Principal Investigator — Brigham and Women's Hospital; John P. Forman, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: VITAL Study website — http://www.vitalstudy.org